CLINICAL TRIAL: NCT00745147
Title: Comparison of Chinese Herbal Formula and Lactulose for Adults With Chronic Constipation-a Randomized ,Double-Blind, Controlled Trial
Brief Title: Comparison of TCM and Laxatives for Adults With Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chien-Hsun Huang, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200803029M
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Constipation
Keywords: constipation; traditional Chinese medicine; Chinese herbal formula; lactulose; cost-effective; long-term care
MeSH Terms: conditions — Constipation | interventions — Lactulose; Laxatives

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Chinese herbal formula + Placebo of duphalac
  Interventions: Drug: Chinese herbal formula (CCH1)
- B (Active Comparator): Duphalac + Placebo of Chinese herbal formula
  Interventions: Drug: Duphalac

INTERVENTIONS:
Drug: Chinese herbal formula (CCH1) — initial dose of 1.5/3.0/4.5gm herbal powder with 15/30/45ml placebo of duphalac, respectively, per day for mild/moderate/severe constipation, then titrated
  Other Names: TCM
  Arms: A
Drug: Duphalac — initial dose of 15/30/45ml duphalac with 1.5/3.0/4.5gm placebo of herbal powder, respectively, per day for mild/moderate/severe constipation, then titrated
  Other Names: Laxative
  Arms: B

SUMMARY:
The purpose of the study is to compare the therapeutic efficacy, safety, cost-effectiveness and maintenance effect between Chinese herbal formula and lactulose on chronic constipation in long-term care.

DETAILED DESCRIPTION:
Although many people regard regular defecation as important factor to maintain healthy, constipation is still a common problem in general population. According to some surveys, constipation affects approximately 50% to 73% of nursing home residents. Because the symptoms cause serious impairment of life quality, laxatives are commonly prescribed for people and over-prescribing of laxatives is also common. Despite the large sums spent on laxatives, there have been few advances in laxative treatment in the last 50 years and there have been minimal research addressing the problem. Therefore constipation was labeled as "the neglected symptoms".

There is unsatisfactory effect by currently pharmacologic therapies and preventive strategies for constipation. Contrarily, they had abundant clinical experiences and medical records for constipation in traditional Chinese medicine. So we follow the worldly trend to do the research of integrative Chinese medicine and Western medicine since WHO launched the first global strategy on traditional and complementary/alternative medicine (TM/CAM) to assist countries to create a stronger evidence base of the TM/CAM products and practices.

The study will be performed under randomized, double-blind, placebo controlled, parallel design. The object of this study is the residents in nursing homes. After intake of Chinese herb, improving constipation and care quality, decreasing the need of enema or digital maneuver, minimizing the dosage of rescue laxatives and saving the medical expenditure will be expected.

ELIGIBILITY:
Inclusion Criteria:

* men and non-pregnant women who are at least 20 years of age
* patients who have been adequately informed of the nature and risks of the study and who have given written informed consent prior to receiving study medication
* the one who meet any one of the following three criteria: 1.RomeIII criteria; 2.at least once a week of enema/suppository use/digital maneuver in past three months; 3.laxative use in more than half time of last three months

Exclusion Criteria:

* known severe renal or hepatic insufficiency,
* known colorectal cancer, anal abscess, anal fistula, anal fissure, rectocele, inflammatory bowel diseases, or gastrointestinal obstruction;
* unknown cause of gastrointestinal bleeding or acute infection
* neuromuscular dystrophy or spinal cord injury induced constipation
* history of drug abuser
* unstable psychiatric disorders
* women who are pregnant, as determined by a urine pregnancy test
* use of an investigational drug (within 30days prior to enrolled)
* known allergies to the component of study medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
frequency of spontaneous bowel movement | every week

SECONDARY OUTCOMES:
amount of rescue laxative use | every week
stool consistency | every week
stool amount | every week
global assessment of efficacy | 2 months
safety evaluation | every week
frequency of enema/suppository use/digital maneuver | every week
medical cost per spontaneous bowel movement | every week

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsun Huang, MD, MSc, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Yun-Lin Branch, Douliu, Yun-Lin, Taiwan

REFERENCES:
- [Background] Lembo A, Camilleri M. Chronic constipation. N Engl J Med. 2003 Oct 2;349(14):1360-8. doi: 10.1056/NEJMra020995. No abstract available. PMID 14523145